CLINICAL TRIAL: NCT00900744
Title: A Pilot Study of Varying Doses of Tamoxifen in the Setting of Genetic Polymorphisms of CYP2D6
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 08-1373; IF#1248430; HSM10-00403
Record Dates: First submitted 2009-05-11; First posted 2009-05-13 (Estimated); Last update posted 2017-08-25 (Actual); Status verified 2017-08

CONDITIONS: Breast Cancer
Keywords: Tamoxifen; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tamoxifen: 20mg daily
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — 20 mg daily
  Other Names: Nolvadex®

SUMMARY:
The investigators plan to examine endoxifen and 4-OH-Tam as a function of the tamoxifen dose in patients with a genetic CYP2D6 polymorphism. The investigators also plan to investigate other genetic variations in the metabolism of tamoxifen.

DETAILED DESCRIPTION:
Endocrine therapy has proven to be an extremely effective therapy in breast cancer. For women with hormone-receptor-positive tumors, tamoxifen given for as little as two years results in a statistically significant recurrence and survival benefit. The benefits increase as the duration of treatment increase, up to 5 years, so that among women treated for five years, tamoxifen can result in up to a 46 percent annual reduction in the recurrence rate and up to a 28 percent annual reduction in the death rate. This means that about half of the recurrences and more than one fourth of the deaths each year are prevented by tamoxifen treatment. However, despite initial successful responses, many patients on tamoxifen relapse and die from progressive disease. Consequently, tamoxifen resistance remains a major clinical problem in the management of breast cancer.

Tamoxifen is metabolized by cytochrome P450 2D6 (CYP2D6) to the more potent metabolites 4-hydroxy-tamoxifen (4-OH-TAM) and 4-hydroxy-N-desmethyltamoxifen (endoxifen). Variations in the metabolic capacity of this enzyme have shown to be an independent predictor of breast cancer relapse and death. To date, studies have not correlated tamoxifen doses to CYP2D6 genotype status or associated tamoxifen doses to endoxifen and 4-OH-tamoxifen.

The investigators plan to examine endoxifen and 4-OH-Tam as a function of the tamoxifen dose in patients with a genetic CYP2D6 polymorphism. The investigators also plan to investigate other genetic variations in the metabolism of tamoxifen. The possible identification of gene variants that alter tamoxifen's metabolism may improve initial dose selection and therefore optimize treatment outcome in the future.

In addition to examining polymorphisms in CYP2D6, other genes will be examine that may influence the metabolism of medications.

ELIGIBILITY:
Inclusion Criteria:

* Women taking tamoxifen 20mg a day
* Tamoxifen use for > 90 days.
* Use an accepted barrier form of contraception.

Exclusion Criteria:

* Patients are excluded if they are pregnant or lactating; if pre- menopausal, the patient will have a documented negative pregnancy test and use an accepted barrier form of contraception.
* Patients are excluded if they have a medical history of Hepatitis B. Hepatitis C or HIV
* Patients are excluded if they use Tobacco
* Patients are excluded if they have a medical history of hereditary hemochromatosis
* Patients are excluded if they have elevated AST (SGOT), ALT (SGPT), Bilirubin or Alkaline Phosphate

  o Defined as greater than 2 1/2 times the upper limit of normal
* Patients are excluded if they are being treated with chemotherapy
* Patients are excluded if they are taking any of the following oral medications, as they are potent CYP2D6 inhibitors:

  * Fluoxetine (Prozac)
  * Miconazole (Monistat)
  * Paroxetine (Paxil)
  * Quinidine
  * Ritonavir (Norvir)
  * Atorvastatin (Lipitor)
  * Carvedilol (Coreg)
  * Clarithromycin (Biaxin)
  * Dipyridamole (Persantine)
  * Erythromycin
  * Grapefruit Juice
  * Itraconazole (Sporanox)
  * Ketoconazole
  * Mefloquine
  * Nelfinavir (Viracept)
  * Nicardipine (Cardene)
  * Nilotinib
  * Propranolol (Inderal)
  * Ranolazine (Ranexa)
  * Saquinavir ( Invirase)
  * Verapamil Covera-HS
  * Warfarin (Coumadin)
  * Chlorpromazine (Thorazine)
  * Cinacalcet (Sensipar)
  * Delavirdine (Rescriptor)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a genetic CYP2D6 polymorphism
Sampling Method: Non-Probability Sample
Enrollment: 121 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Specific human 2D6 variants measurement(s) or observation(s) | every two weeks

CONTACTS AND LOCATIONS:
Overall Officials: George Raptis, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States